CLINICAL TRIAL: NCT04817059
Title: The Impact of Customized Head Molds on Motion and Motion-related Artifacts From Structural and Functional MRI Scans in Children
Brief Title: Reducing Head Motion With Customized Head Mold in Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Robust Motion
Record Dates: First submitted 2021-03-23; First posted 2021-03-25 (Actual); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Child Development; Adhd; Neuroimag
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Head mold on (Experimental)
  Interventions: Device: Caseforge headcase
- Head mold off (No Intervention)

INTERVENTIONS:
Device: Caseforge headcase — We used a custom-fitted styrofoam head mold designed to reduce head motion during MRI scanning.
  Arms: Head mold on

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a customized head mold for reducing head motion during MRI scanning in young children.

DETAILED DESCRIPTION:
Each participant completed a dedicated session for mock scanning before we acquired two sets of sMRI and fMRI scans. One scan set was collected using the head mold and the other without, and the scans were counterbalanced in order across participants. Using a specialized sMRI sequence embedded with vNAVs, we directly measured head motion during sMRI in order to more accurately evaluate the head mold's impact on structural metrics. To evaluate the feasibility and tolerability of the head mold, we concluded the scanning sessions with a brief interview that gauged participants' scanning experience and tolerance of the head mold. We investigated whether head molds would reduce head motion compared to standard scanning procedures and whether those reductions would result in improved data quality. We also tested the extent to which reductions in head motion impacted estimations of cortical volume and functional connectivity. Prior to data collection, we evaluated the noise dosage levels of the head mold condition, given the limited space available for additional hearing protection devices in the head coil while the head mold is on. We also assessed whether the head molds could balance head motion between typical and ADHD populations, and whether clinical variables such as ADHD diagnosis and trait anxiety, as determined by parent-reported dimensional measures, can predict head mold efficacy.

ELIGIBILITY:
Inclusion Criteria:

* between ages 5 - 10
* ADHD diagnosis as determined by parent self-report

Exclusion Criteria:

* no MRI contraindications and no history of head injuries or seizures.

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2019-08-08 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Head motion during MRI scanning | during MRI scanning
  Head motion during MRI scanning was estimated and compared with and without the head mold on.

SECONDARY OUTCOMES:
Image quality | during MRI scanning
  MRI quality was also compared between experimental and control conditions.

CONTACTS AND LOCATIONS:
Overall Officials: Cameron Craddock, PhD, Principal Investigator — University of Texas at Austin
Locations (1):
- Health Discovery Building Biomedical Imaging Center, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
All data will be de-identified using standards conforming to HIPAA guidelines. Consistent with the model setup by the International Data Sharing Initiative (INDI) effort, data will be distributed via the NITRC-based Functional Connectome Project (FCP)/INDI website (http://fcon_1000.projects.nitrc.org/). The following steps will be carried out to ensure that no identifying or protected health information is released:
  * All imaging files will be stripped of fields containing protected health information, and date of exam will be removed
  * Anatomical images will have face information removed or obscured.
  * Random ID numbers will be generated and assigned to each dataset prior to release.
  Legal guardians of the child participants will be asked if they consent to having their data shared publicly, as well as privately with other University of Texas at Austin researchers. If they do not consent to having their data shared, they may still participate in the study without penalty.
Supporting Information: Study Protocol